CLINICAL TRIAL: NCT03978078
Title: Development of a Prospective Clinicobiological Database in Metastatic Digestive Cancers
Brief Title: A Clinicobiological Database in Metastatic Digestive Cancers
Acronym: BCB-CBIO-DIG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICM-URC 2016/08
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Digestive System Neoplasm
Keywords: colorectal; pancreas; stomach; oesophagus; bile duct; small intestine; cancer
MeSH Terms: conditions — Digestive System Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): For all the patients include in the study :
  - Blood samples collected at different times : Before treatment, during treatment (approximately every other month) through the end of treatment
  In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — - Blood samples collected at different times : Before treatment, during treatment (approximately every other month) through the end of treatment

SUMMARY:
Creation of a collection of blood samples that will be collected before and then under treatment in patients with digestive adenocarcinoma during the 1st and 2nd metastatic line and which, depending on scientific progress, can be used for research projects aimed at developing tailored patient management strategies.

DETAILED DESCRIPTION:
Digestive cancers account for 30% of all cancers. The most common of these colorectal cancer (CRC) is the third most common cause of cancer in the world.

In the metastatic phase, patients with digestive cancers generally benefit from medical treatment based on cytotoxic chemotherapy, which can be combined with targeted therapy in certain locations. Their use is based on demonstrating a significant improvement in the overall survival of patients.

However, the therapeutic choice and follow-up of these treatments as a the first line treatment and beyond remain difficult given a cruel lack of biomarkers capable of predicting the response to these different molecules upstream but also usable during treatment to evaluate their efficacy or identify the development of secondary resistance mechanisms.

Indeed, the only biomarkers currently validated and used before the initiation of anti-cancer treatment to stratify patients are:

* the search for mutations in Kirsten rat sarcoma viral oncogene homolog (KRAS) and neuroblastoma rat sarcoma viral oncogene (NRAS) oncogenes as predictive factors for non-response to anti-Epidermal Growth Factor receptor (EGFR) in colorectal adenocarcinomas.
* the search for overexpression of the human epidermal growth factor (HER2) receptor to introduce trastuzumab treatment in esophageal adenocarcinomas.

In addition, they are conventionally determined from tumor tissue, which requires an invasive biopsy or surgical sampling that is difficult to repeat over time.

In this context, it seems essential to us to identify new parameters allowing a better personalization of anti-cancer treatments, by favouring blood biomarkers that have the advantage of being evaluated in a minimally invasive manner and therefore be repeated to be able to judge tumor dynamics.

To this end, we propose the creation of a collection of samples that will be collected before and then under treatment in patients with digestive adenocarcinoma in the 1st and 2nd metastatic line and which, depending on scientific progress, can be used for research projects aimed at developing tailored patient management strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old
2. Histological documentation of adenocarcinoma of the colon or rectum, small intestine, pancreas, stomach, bile duct, oesophagus
3. Patient who will receive a first or second line metastatic chemotherapy and/or targeted therapy
4. Informed consent form (ICF) signed

Exclusion Criteria:

1. Male or female < 18 years old
2. Non-adenocarcinoma histological type
3. Patient already undergoing specific treatment (chemotherapy and/or targeted therapy) in 1st or 2nd metastatic line
4. Pregnant and/or breastfeeding woman
5. Patient not affiliated to a social security system
6. Patient whose regular follow-up is impossible for psychological, family, social or geographical reasons
7. Patient who is included in a Phase I-II therapeutic trial modifying usual management and involving additional and specific blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Number of clinical risk factors for metastatic digestive cancer | Until the study completion : 54 months
Number of biological risk factors for metastatic digestive cancer | Until the study completion : 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Thibault Mazard, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (1):
- Institut régional du cancer de Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ren JS, Masuyer E, Ferlay J. Global estimates of cancer prevalence for 27 sites in the adult population in 2008. Int J Cancer. 2013 Mar 1;132(5):1133-45. doi: 10.1002/ijc.27711. Epub 2012 Jul 26. PMID 22752881
- [Background] Karapetis CS, Khambata-Ford S, Jonker DJ, O'Callaghan CJ, Tu D, Tebbutt NC, Simes RJ, Chalchal H, Shapiro JD, Robitaille S, Price TJ, Shepherd L, Au HJ, Langer C, Moore MJ, Zalcberg JR. K-ras mutations and benefit from cetuximab in advanced colorectal cancer. N Engl J Med. 2008 Oct 23;359(17):1757-65. doi: 10.1056/NEJMoa0804385. PMID 18946061
- [Background] Douillard JY, Oliner KS, Siena S, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Williams R, Rong A, Wiezorek J, Sidhu R, Patterson SD. Panitumumab-FOLFOX4 treatment and RAS mutations in colorectal cancer. N Engl J Med. 2013 Sep 12;369(11):1023-34. doi: 10.1056/NEJMoa1305275. PMID 24024839
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210